CLINICAL TRIAL: NCT02778932
Title: Comparison of Immobilization Quality During General Anesthesia for Pars Plana-vitrectomy With and Without Neuromuscular Blockade and Endotracheal Intubation Measured by a Questionnaire
Brief Title: Comparison of Intubation and Laryngeal Mask for Pars Plana Vitrectomy
Acronym: ITNLMAPPV
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Studienleiter, University Hospital Schleswig-Holstein
Other Study IDs: D 466/16
Record Dates: First submitted 2016-05-08; First posted 2016-05-20 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Muscle Relaxation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intubation: General anesthesia including intubation and muscle relaxation
- Laryngeal Mask: General anesthesia including laryngeal mask without muscle relaxation

SUMMARY:
Pars plana vitrectomy is usually performed under general anesthesia including endotracheal intubation and muscle relaxation. However, for short procedures anesthesia using a laryngeal mask without muscle relaxation is also common in practice. In this observational study the incidence of patient movement will be examined between these anesthesia techniques.

DETAILED DESCRIPTION:
Usually eye surgery can be safely performed under local anesthesia. However, if the eye is opened during the procedure, general anesthesia may be a safer alternative. The intraocular pressure is less stable in wake patients than in anesthetized patients and increasing intraocular pressure can lead to prolapse of vitreous. Moreover, wake patients may move during the procedure and movement during surgery can cause serious lesions of the retina with consecutive loss of vision due to intraocular instruments.

A typical intraocular procedure is vitrectomy. During vitrectomy the vitreous body is removed and substituted by silicon oil or gas. Vitrectomy is usually performed by inserting instruments through the pars plana in the eye. The pars plana, an area between iris and retina, contains no structures essential for vision. On one side of the eye a light source and access for intraocular infusion is introduced into the eye through the pars plana. An infusion is connected and fixed at 60 cm above eye level thus maintaining intraocular pressure by gravity. On the opposite side of the eye instruments like scalpels, scissors or an instrument combining cutting and suction of vitreous can be inserted through a tube. Common indications for vitrectomy are vitreous body bleedings or retinal detachment.

Reliable immobilization by anesthesia is mandatory for vitrectomy. However, anesthesia for vitrectomy is complicated by the fact that the anatomical structures at risk are reached very early during operation and consequently there is not much time to adopt anesthesia dosage to individual patient's needs. At the end of the procedure the critical area is left a few minutes before conjunctival suture leaving a relatively short period of time for recovery from anesthesia until extubation.

Possibly due to these difficulties deviation of vision axis and patient movements are not uncommon during general anesthesia for eye operations. Usually these events can be dealt with by supplementation of anesthesia and muscle relaxation, but they can lead to impairment of operation conditions and put the patient at risk of eye damage and loss of vision. Rossiter and co-workers investigated quality of immobilisation in 52 patients during eye surgery. Even small eye movements like upward deviation of the vision axis have been regarded as incomplete immobilisation in this study because they interfere with surgery and thereby increase the risk of complications.

In four of these 52 patients (7.6 %) eye movements have been observed during surgery (Rossiter 2006). It has been shown by a further study that these deviations can be quantified and depend from the patient's preoperative findings (Daien 2013).

Vitrectomy is performed as 20-gauge- or 23-gauge sutureless transconjunctival vitrectomy, depending of the diameter of the intraocular access channel (Aylward 2011)3. Generally, operation time is considerably shorter for 23-Gauge-vitrectomie, because no conjunctival suture is needed. Hence, 23 Gauge-vitrectomies are performed under general anesthesia using a laryngeal mask without muscle relaxation at our institution. 20-Gauge-vitrectomies are performed under general anesthesia with endotracheal intubation due to longer operation times. However, total muscle relaxation is maintained only during the first 30 - 45 min of surgery until reliable immobilization is reached by volatile anesthetics. The results of Rossiter and co-workers showed that eye movements occurred only during surgery without muscle relaxation in their study. Hence, it may be argued that immobilization by balanced anesthesia only during 23 Gauge-vitrectomy and during the second half of 20 Gauge-vitrectomy may be inferior to immobilization by addition of muscle relaxants.

Objective of this prospective observational study is the comparison of immobilization quality during general anesthesia for pars plana-vitrectomy with and without neuromuscular blockade and endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pars plana vitrectomy under general anesthesia

Exclusion Criteria:

* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing pars plana vitrectomy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Daien V, Turpin C, Lignereux F, Belghobsi R, Le Meur G, Lebranchu P, Pechereau A. Determinants of ocular deviation in esotropic subjects under general anesthesia. J Pediatr Ophthalmol Strabismus. 2013 May-Jun;50(3):155-60. doi: 10.3928/01913913-20130226-01. Epub 2013 Mar 5. PMID 23451722
- [Background] Rossiter JD, Wood M, Lockwood A, Lewis K. Operating conditions for ocular surgery under general anaesthesia: an eccentric problem. Eye (Lond). 2006 Jan;20(1):55-8. doi: 10.1038/sj.eye.6701789. PMID 15650757
- [Background] Spiteri N, Sidaras G, Czanner G, Batterbury M, Kaye SB. Assessing the quality of ophthalmic anesthesia. J Clin Anesth. 2015 Jun;27(4):285-9. doi: 10.1016/j.jclinane.2015.01.008. Epub 2015 Feb 18. PMID 25704674

RESULTS

PARTICIPANT FLOW:
Groups:
- Intubation: Patients receiving general anesthesia including intubation and muscle Relaxation for pars plana-vitrectomy
Period: Overall Study
Arm/Group | Intubation | Laryngeal Mask
Started | 74 | 74
Completed | 74 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ITN and Relaxation: General anesthesia including intubation and muscle relaxation
- LM Without Relaxation: General anesthesia including laryngeal mask without muscle relaxation
- Total: Total of all reporting groups
Arm/Group | ITN and Relaxation | LM Without Relaxation | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 43 | 82
  >=65 years | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12) | 64 (15) | 64 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 37 | 68
  Male | 43 | 37 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 74 | 74 | 148

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Moving During Pars Plana Vitrectomy (Count of Participants)
Description: Movements of patients and abnormal deviations of eye position during surgery were reported to the anesthetist by the surgeon and noted by the anesthetist. Each patient with movement or abnormal deviations of eye position was counted as patient moving during pars plana vitrectomy (Count of participants). No score was used to report movement. Hence, no further score informations can be included.
Time Frame: The estimated period of time over which the event is assessed is the time between incision and suture (estimated period of time: 30 - 180 min).
Population: Patients scheduled for pars plana vitrectomy
Measure: Number; unit: participants
Groups:
- ITN Without Relaxation: General anesthesia including intubation and muscle relaxation
Arm/Group | ITN Without Relaxation | LM Without Relaxation
Number analyzed (Participants) | 74 | 74
participants | 0 | 9

2. Secondary Outcome: Quality of Immobilization
Description: Quality of immobilization will be investigated by interviewing surgeons using a standardized questionnaire including quality of eye position, general immobilization, akinesia of the eye, blood loss, intraocular pressure, surgeon satisfaction with immobilization and anesthesia. Outcome measure is the surgeon's satisfaction measured on a score between 0 and 10 (Score title: Questionnaire for quantification of immobilization during general anesthesia for pars-plana vitrectomy. Higher scores mean a better outcome. 0 = None (Minimum), worst outcome, 10 = Maximal (Maximum), best outcome, Title: Quality of immobilization)
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Groups:
- ITN Without Relaxation: General anesthesia including intubation and muscle Relaxation
  Result: Surgeon's satisfaction was 10 [0-10] (Median [Range], Rating Scala: 0 (none) to 10 (maximal))
- LM Without Relaxation: General anesthesia including laryngeal mask without muscle Relaxation
  Result: Surgeon's satisfaction was 10 [0-10] (Median [Range], Rating Scala: 0 (none) to 10 (maximal))
Arm/Group | ITN Without Relaxation | LM Without Relaxation
Number analyzed (Participants) | 74 | 74
score on a scale | 10 [8 to 10] | 10 [8 to 10]

ADVERSE EVENTS:
Time Frame: The time period over wich adverse event data were collected was 7 months.
Groups:
- ITN With Relaxation: General anesthesia including intubation and muscle relaxation
Arm/Group | LM Without Relaxation | ITN With Relaxation
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/74
Other Adverse Events (participants affected / at risk) | 0/74 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes